CLINICAL TRIAL: NCT04974229
Title: Sensory Profiles as Predictors of Central Sensitization in Low Back Pain: A Prospective Cohort Study.
Brief Title: Prognostic Factor Research of Sensory Profiles in Development of Central Sensitization
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Pieter Graper, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: ProgCohSt-M15.169564
Record Dates: First submitted 2021-07-06; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Sensory Profiles; Central Sensitisation; Low Back Pain; Nociplastic Pain
Keywords: Prognostic factors research; Sensory Profiles; Central Sensitisation; Low back pain; Nociplastic Pain
MeSH Terms: conditions — Low Back Pain; Nociplastic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — patients with acute low back pain (< 6 weeks) were consecutively included with or without radiating pain, aged 18 to 60 years with a pain-free episode for at least 3 months before the onset of their current back pain. They were also required to be able to read and understand the Dutch language.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute non-specific low back pain: patients with acute low back pain of (< 6 weeks) were consecutively included with or without radiating pain, aged 18 to 60 years with a pain-free episode for at least 3 months before the onset of their current back pain. They were also required to be able to read and understand the Dutch language.
  Interventions: Other: In line with the Dutch guideline for non-specific low back pain, Standard usual care for non-specific low back pain was applied.

INTERVENTIONS:
Other: In line with the Dutch guideline for non-specific low back pain, Standard usual care for non-specific low back pain was applied. — In line with the Dutch guideline for non-specific low back pain, Standard usual care or non-specific low back pain was applied.
  Other Names: In line with the Dutch guideline for low back pain, Standard usual care or non-specific low back pain was applied.

SUMMARY:
A longitudinal observational cohort study to investigate the value of prognostic factors, here sensory profiles , and others, in the development of central sensitization in the low back pain population. A type 2 prognostic factor research following the PROGRESS framework. Sensory profiles are identified a prognostic factors which can predict the development of central sensitization in the low back pain population.

DETAILED DESCRIPTION:
After performing an univariable linear regression analyses the regression model predicts the dependent variable, central sensitization, significantly, and the models are significant prediction factors of the development of central sensitization. In unadjusted analyses, all four sensory profiles were significantly associated with the development of central sensitization (P<0.001).

After adjusting for pain, disability, age, and duration of low back pain, baseline sensory profiles remained significant predictors of central sensitization. On the other hand, all other predictor variables did not contribute to the prediction of central sensitization.

ELIGIBILITY:
Inclusion Criteria:

* acute low back pain (< 6 weeks)
* with or without radiating pain
* aged 18 to 60 years
* a pain-free episode for at least 3 months before the onset of their current back pain
* read and understand the Dutch language.

Exclusion Criteria:

* previous lumbar spinal surgery
* lumbar radicular syndrome
* specific cause of low back pain
* lumbar spinal stenosis
* current malignancy
* spondyloarthropathy
* osteoporosis
* spondylolisthesis
* major trauma
* infection
* systemic disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants were recruited primary care physiotherapy practices randomly spread throughout the Netherlands. Participants with acute low back pain were consecutively included by physiotherapists.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory score | 12 weeks
  The validated questionnaire Central Sensitization Inventory which scores on a 5 point scale ranging from 0-100. A higher score indicated a higher degree of central sensitization.
Adolescent/Adult Sensory Profile score | 0 weeks
  Adolescent/Adult Sensory Profile measures 4 sensory profiles (sensation avoiding, sensation sensitive, sensation seeking, low registration) on ad 5 point scale, and is validated in the low back pain population. Scores range from 15-60 points per variable. A higher score means a higher degree of sensitivity for the specific sensory profile.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale score | Baseline (0 weeks)
  Numeric Pain Rating Scale measures experienced level of pain, which consist of one question ranging van 0 (no pain)-10 (most extreme pain imaginable).
Pain Disability Index score | Baseline (0 weeks)
  The Pain Disability Index evaluates the effect on seven life-related domains. Each domain is measured by 1 question, with a total of 7 questions, on an 11 point scale, from 0 (no disability) to 10 (completely disabled). Previously established reliability and internal consistency are acceptable in patients with chronic pain.
age | Baseline (0 weeks)
  The included age (years) ranged from 18-60 score. A higher age indicates a worse prognoses of low back pain.
duration of low back pain | Baseline (0 weeks)
  Duration of low back pain was assessed in weeks. The included duration of low back pain ranged from 0-6 weeks. A longer duration is not better or worse.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Scafoglieri, PhD, Study Director — VUB
Locations (1):
- Vrije universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No